CLINICAL TRIAL: NCT05322564
Title: Standardization of Post-operative Opiate Prescriptions for Same-day Ankle and Wrist Fracture Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Ottawa Hospital (Other)
Responsible Party: Principal Investigator, Zoe Rubin, Surgical Resident, The Ottawa Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: Post-op opiate standardization
Record Dates: First submitted 2022-02-09; First posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Opioid Use; Post-operative Pain; Prescription Opioid Abuse; Fracture, Ankle; Fracture Wrist; Surgery
MeSH Terms: conditions — Pain, Postoperative; Opioid-Related Disorders; Ankle Fractures; Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care cohort (No Intervention): Eligible wrist and ankle fracture patients booked for open reduction and internal fixation through our emergency day surgery program will be recruited and consented via telephone prior to their surgery date. The study participants will receive a post-operative prescription at the discretion of their attending surgeon, fellow or resident, with no intervention from the researchers involved in this study. On post-operative day three and post-operative day ten, these patients will be contacted by phone by the research team and asked to respond verbally to a questionnaire. Measures including quantity of opiates consumed, pain intensity and satisfaction with pain treatment will be recorded.
- Standardized prescription cohort (Experimental): Using the data collected from the standard of care cohort, a standardized pain prescription will be created. The average quantity of opiates consumed by the standard of care participants will be used to guide the quantity of opiates to be prescribed on the standardized prescription. In this arm, all eligible patients will be contacted and recruited by telephone prior to their surgery. These patients will be flagged on the day of surgery and given the standardized prescription post-operatively. They will then be asked to respond to the same questionnaires as the standard of care cohort via telephone on post-op day three and post-op day ten.
  Interventions: Other: Standardized opiate prescription

INTERVENTIONS:
Other: Standardized opiate prescription — The standardized prescription will include a single opiate, with a fixed dose and number of tablets. It will also include non-opiate adjuncts commonly prescribed at our institution, namely acetaminophen and an anti-inflammatory medication.
  Arms: Standardized prescription cohort

SUMMARY:
The purpose of this prospective cohort study is to evaluate the opiate prescribing patterns post open reduction and internal fixation (ORIF) of wrist and ankle fractures at the Ottawa Hospital.

The primary objective would be to examine the quantity and duration of opiates consumed by the study population, as well as the participant's overall satisfaction with pain control. the investigators will assess whether there is a discrepancy between the quantity of pills prescribed and what is being consumed.

With the data collected, the secondary objective would be to create a standardized pain prescription, which the investigators would implement in the second phase of this prospective study. Opiate pills consumed, pain satisfaction and left-over narcotics would again be assessed.

The overall goal of this study is to produce an appropriate standardized post-operative prescription, where the number of opiates prescribed mirrors what is being consumed. This would cut down on the quantity of left-over narcotics, helping to reduce the incidence of opiate dependency and diversion in the Ottawa community.

DETAILED DESCRIPTION:
This is a multiphase study that will begin with a retrospective review of the prescribing patterns at the Ottawa Hospital. The post-operative prescriptions of 50 wrist fracture and 50 ankle fracture patients booked for same day fracture fixation will be reviewed. The type and quantity of opiate pills prescribed, as well as the other multimodal analgesics prescribed will be collected. Phase one will provide the investigators with data regarding the recent prescribing trends at the Ottawa Hospital prior to beginning the prospective phase of the study.

Phase two and three of the study involves collecting data from two prospectively collected cohorts - the standard of care cohort (phase 2) and the standardized prescription cohort (phase 3).

In phase two, eligible wrist and ankle fracture patients booked for open reduction and internal fixation through the Walking Wounded (emergency day surgery) program will be recruited and consented via telephone prior to their surgery date. The study participants will receive a post-operative prescription at the discretion of their attending surgeon, fellow or resident, with no intervention from the researchers involved in this study. On post-operative day three and post-operative day ten, these patients will be contacted by phone by the research team and asked to respond verbally to a questionnaire that will record the following measures - quantity of opiates consumed/left-over, pain intensity, satisfaction with pain treatment and other non-opiate medications taken.

Using the data collected from phase two, a standardized pain prescription will be created. The average quantity of opiates consumed by the phase two participants will be used to guide the quantity of opiates to be prescribed on the standardized prescription. Similar to recruitment in phase two, in phase three, all eligible patients will be contacted and recruited by telephone prior to their surgery. These patients will be flagged on the day of surgery and given the standardized prescription post-operatively. They will then be asked to respond to the same questionnaires via telephone on post-op day three and post-op day ten.

ELIGIBILITY:
Inclusion Criteria:

* Ankle and wrist fracture patients booked for ORIF (via Walking Wounded program)
* Opioid naïve (Opiates prescribed in emergency not included)
* Competent to give informed consent and respond to questionnaires independently
* English or French speaking

Exclusion Criteria:

* Admission to hospital pre- or post-operatively
* Chronic opioid use for pain unrelated to injury
* Chronic pain in injured extremity, unrelated to acute injury
* Previous fracture/surgery to injured limb
* Revision ORIF
* Dementia or cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Patient reported pain satisfaction | Measures will be recorded on days 3 postoperatively
  Patient reported pain satisfaction between those receiving standard of care, and those receiving the novel standardized prescription will be compared. Treatment satisfaction will be measured using the 11-point ordinal rating of pain intensity (numeric rating scale) and an 11-point ordinal rating of satisfaction with pain relief. In addition to the numerical rating scale, A verbal rating scale (VRS), will also be used to qualify pain control. The VRS consists of a list of descriptors that represent varying degrees of pain intensity. Each of these descriptors has a number associated with it (e.g., 0 = none, 1 = mild pain, 2 = moderate pain, 3 = severe pain, and 4 = intolerable pain). Comparable to the VRS, the Likert scale will similarly be used to qualify treatment satisfaction (e.g., 0 = Very satisfied, 1 = somewhat satisfied, 2 = neither satisfied nor dissatisfied, 3 = somewhat dissatisfied, and 4 = very dissatisfied).
Patient reported pain satisfaction | Measures will be recorded on day 10 postoperatively
  Patient reported pain satisfaction between those receiving standard of care, and those receiving the novel standardized prescription will be compared. Treatment satisfaction will be measured using the 11-point ordinal rating of pain intensity (numeric rating scale) and an 11-point ordinal rating of satisfaction with pain relief. In addition to the numerical rating scale, A verbal rating scale (VRS), will also be used to qualify pain control. The VRS consists of a list of descriptors that represent varying degrees of pain intensity. Each of these descriptors has a number associated with it (e.g., 0 = none, 1 = mild pain, 2 = moderate pain, 3 = severe pain, and 4 = intolerable pain). Comparable to the VRS, the Likert scale will similarly be used to qualify treatment satisfaction (e.g., 0 = Very satisfied, 1 = somewhat satisfied, 2 = neither satisfied nor dissatisfied, 3 = somewhat dissatisfied, and 4 = very dissatisfied).

SECONDARY OUTCOMES:
Average quantity of opioids prescribed in the standard of care cohort measured using morphine equivalents. | Prescription information will be collected at a single point prior to post-operative day 3.
  The quantity of opioids prescribed per patient will be converted to Morphine Milligram Equivalents (MME). Data on quantity and types of opiates prescribed, as well as other non-opiate adjuncts, will be collected through EPIC, our institution's electronic health records system.
Average quantity of opioids consumed post-operatively in both cohorts | Measures will be recorded on day 3 postoperatively
  The quantity of opiates consumed per patient will be collected on post-operative day three, by asking the study participant to count the number of pills remaining in their opiate prescription bottle.
Average quantity of opioids consumed post-operatively in both cohorts | Measures will be recorded on day 10 postoperatively
  The quantity of opiates consumed per patient will be collected on post-operative day ten, by asking the study participant to count the number of pills remaining in their opiate prescription bottle.
Average quantity of left-over/unused opiates | Post-operative day 10
  The quantity of opiates remaining per patient will be collected on post-operative day ten, by asking the study participant to count the number of pills remaining in their opiate prescription bottle.
Distribution of use of different opioids and non-opioid adjuncts prescribed | Prescription information will be collected at a single point prior to post-operative day 3.
  The variety of different opiate molecules and non-opiate adjuncts prescribed will be collected and the frequency that each type is being used at our institution will be analyzed.
The difference in consumption patterns between patients receiving peripheral nerve blocks versus those who haven't received a regional anesthetic. | Measures will be recorded on days 3 postoperatively
  Average quantity of opioids consumed post-operatively will be compared between the patients receiving peripheral nerve blocks versus those who haven't received a regional anesthetic.
The difference in consumption patterns between patients receiving peripheral nerve blocks versus those who haven't received a regional anesthetic. | Measures will be recorded on day 10 postoperatively
  Average quantity of opioids consumed post-operatively will be compared between the patients receiving peripheral nerve blocks versus those who haven't received a regional anesthetic.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sabatino MJ, Kunkel ST, Ramkumar DB, Keeney BJ, Jevsevar DS. Excess Opioid Medication and Variation in Prescribing Patterns Following Common Orthopaedic Procedures. J Bone Joint Surg Am. 2018 Feb 7;100(3):180-188. doi: 10.2106/JBJS.17.00672. PMID 29406338
- [Background] Saini S, McDonald EL, Shakked R, Nicholson K, Rogero R, Chapter M, Winters BS, Pedowitz DI, Raikin SM, Daniel JN. Prospective Evaluation of Utilization Patterns and Prescribing Guidelines of Opioid Consumption Following Orthopedic Foot and Ankle Surgery. Foot Ankle Int. 2018 Nov;39(11):1257-1265. doi: 10.1177/1071100718790243. Epub 2018 Aug 19. PMID 30124084
- [Background] Helmerhorst GTT, Zwiers R, Ring D, Kloen P. Pain Relief After Operative Treatment of an Extremity Fracture: A Noninferiority Randomized Controlled Trial. J Bone Joint Surg Am. 2017 Nov 15;99(22):1908-1915. doi: 10.2106/JBJS.17.00149. PMID 29135664
- [Background] Bhashyam AR, Basilico M, Weaver MJ, Harris MB, Heng M. Using Historical Variation in Opioid Prescribing Immediately After Fracture Surgery to Guide Maximum Initial Prescriptions. J Orthop Trauma. 2019 Apr;33(4):e131-e136. doi: 10.1097/BOT.0000000000001392. PMID 30570619
- [Background] Adalbert JR, Ilyas AM. Implementing Prescribing Guidelines for Upper Extremity Orthopedic Procedures: A Prospective Analysis of Postoperative Opioid Consumption and Satisfaction. Hand (N Y). 2021 Jul;16(4):491-497. doi: 10.1177/1558944719867122. Epub 2019 Aug 23. PMID 31441326
- [Background] Kim N, Matzon JL, Abboudi J, Jones C, Kirkpatrick W, Leinberry CF, Liss FE, Lutsky KF, Wang ML, Maltenfort M, Ilyas AM. A Prospective Evaluation of Opioid Utilization After Upper-Extremity Surgical Procedures: Identifying Consumption Patterns and Determining Prescribing Guidelines. J Bone Joint Surg Am. 2016 Oct 19;98(20):e89. doi: 10.2106/JBJS.15.00614. PMID 27869630